CLINICAL TRIAL: NCT04868084
Title: Early Years Physical Activity and Movement Skills Intervention - Feasibility Study to Evaluate an Existing Training Programme for Early Years Practitioners
Brief Title: Early Years Physical Activity and Movement Skills Intervention: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: University of Huddersfield (Other); Teesside University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Early years physical activity
Record Dates: First submitted 2021-03-15; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-02

CONDITIONS: Child Obesity; Activity, Motor; Physical Activity
Keywords: Practitioner; Fundamental movement skills; Educational training; Early years; Preschool
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Non-randomised before and after pilot feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Physical Literacy in the early years. The intervention was delivered by an external provider and designed to provide nursery teachers, teaching assistants and others working with children under age five the knowledge, skills and confidence to deliver enjoyable and engaging lessons which focus on the development of core "fundamental" skills. The course was developed in conjunction with leading Physical Education (PE) consultants, Sports Scientists and Office for Standards in Education, Children's Services and Skills (Ofsted) advisors which covered both the theory about FMS and physical literacy, and practical demonstrations of age-appropriate ways to teach and develop FMS. Staff from the Intervention settings received the six-hour training session. After the training session, school nurseries which were encouraged to speak with the training provider to follow-up the understanding of the training and provide additional help for implementation of the practice learned.
  Interventions: Behavioral: Physical literacy in the early years
- Control (No Intervention): The control nurseries followed their usual practice.

INTERVENTIONS:
Behavioral: Physical literacy in the early years — Intervention nurseries received a 6-hour training session, covering the theory about FMS and practical demonstrations of age-appropriate ways to teach and develop FMS.
  Arms: Intervention group

SUMMARY:
This project aims to test the feasibility of using an existing training course for nursery practitioners (those that care for children aged under 5 years) to improve their ability and confidence to teach fundamental movement skills to the children they care for. 'Fundamental movement skills', or FMS, are based on agility, balance and coordination, and include jumping, throwing, catching, striking and running and are vital for children's involvement in, and enjoyment from, physical activities and sports. The intervention consists of a one-day course given by specialist providers, specifically for those who work with children under 5. The intervention aims to increase practitioner knowledge and awareness, and increase confidence in their ability to provide age-appropriate guidance and settings for FMS and active play. The implication from the training is that the children's FMS and overall physical activity will increase, whilst decreasing time spent in sedentary behaviours. A long-term aim of the project would be the maintenance of a healthy weight by the children and increase in self-efficacy for physical activity. The benefits of the study, therefore, are an increase in practitioner confidence and knowledge, and a positive change in their behaviour during their everyday practice. As this is a feasibility study, the main objective is whether a full trial would be feasible. The primary outcomes are therefore 1. Recruitment (ratio of consented participants to potentially eligible participants approached) 2. Numbers completing study 3. Numbers completing study questionnaires 4. Acceptability of the intervention to participants.

DETAILED DESCRIPTION:
This is a pilot non-randomised controlled trial. The study was approved by the Newcastle University Research Ethics Committee (application number:01223/9764/2016). The intervention consists of a one-day course given by specialist providers, specifically for those who work with children under 5. The training consisted on helping practitioners around fundamental movement skills (balancing, jumping throwing, catching kicking) and helping them to develop a better understanding about the importance of physical activity for early years. The training also covered an introduction to the United Kingdom (UK) physical activity guidelines and how practitioners could translate the physical activity guidelines into practice. The course used an ecological model approach in the delivery of the intervention. The programme provided ideas for: creating enabling environments for physical activity; planning physical activity for all stages of development; balance child-initiated and adult-led physical activities; encourage parent and carer support and promotion of physical activity beyond the nursery setting. Data collection took place between February 2017 and June 2018. All nurseries and schools with nurseries in the Middlesbrough area were eligible to participate and were invited to take part.

The following measures were intended to be collected pre-intervention and 6 months post-intervention (follow-up). Practitioner behaviour was assessed by direct observation adapted from the Communication Supporting Classroom Observation Tool. Each observation lasted approximately 30 min and was conducted by one of the researchers. Knowledge of the physical activity guidelines and benefits of physical activity for early years was assessed by a customised questionnaire. Intentions for behaviour change was assessed by a questionnaire which covered the following domains: Knowledge; Skills; Social/Professional Role & Identity; Belief about Capabilities; Optimism; Beliefs about Consequences; Intentions; Goals- Action Planning; Goals - Priorities; Memory, Attention & Decision Processes; Environmental Context & Resources; Social Influences; Emotion; Behavioural Regulation; Social & Professional Role; Work Environment. Children. Physical activity was measured directly using a thigh-mounted accelerometer (activPAL) which has been validated in young children. Time in sitting, standing and stepping postures was measured during school or nurseries hours. Data were recorded in 15 s epoch and reduced to the percentage of wear time in each of the postures, to account for potential differences in wear time within and between participants. Height (to 0.1cm) and weight (to 0.1kg) were measured twice without socks or shoes, in indoor clothing. BMI was then derived, and z -scores created relative to UK 1990 data. Fundamental movement skills were assessed with the Movement Assessment Battery for Children 2 (Movement ABC-2) which covers fine and gross motor tasks, manual dexterity and balance. Process evaluation. Using focus groups, interviews and a questionnaire with all stakeholders explored the reasons for participation/non-participation of practitioners and families; participants' views and perceptions of the intervention in terms of acceptability, feasibility and usability. All data were exported to SPSS for analyses. Descriptive statistics for all variables of interest were generated

ELIGIBILITY:
Inclusion Criteria:

* Children who are 3 to 4 years old at the time of data collection.
* Children who received parent/guardian consent.
* Children who provided assent to take part in the study.

Exclusion Criteria:

* None

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in fundamental motor skills (FMS) | Baseline and 6 months post-intervention
  FMS, assessed with the Movement Assessment Battery for Children-2 which covers fine and gross motor tasks, manual dexterity and balance. Standard scores are translated to reference percentiles. Low percentiles indicate movement difficulties.
Change in children's physical activity | Baseline and 6 months post-intervention
  Children's physical activity was measured directly using a thigh-mounted accelerometer (ActivPAL) for 7 days

SECONDARY OUTCOMES:
Change in body mass index z-score | Baseline and 6 months post-intervention
  Height (to 0.1cm) and weight (to 0.1kg) were measured twice without socks or shoes, in indoor clothing. BMI was then derived, and z -scores created relative to UK1990 data
Change in practitioner behaviour | Baseline and 6 months post-intervention
  Practitioner behaviour was assessed by direct observation adapted from the Communication Supporting Classroom Observation Tool from the communication trust. Each observation lasted approximately 30 min and was conducted by one of the researchers.
Change in knowledge of the physical activity guidelines | Baseline and 6 months post-intervention
  Knowledge of the physical activity guidelines and benefits of physical activity for early years was assessed by a customised questionnaire
Change in intentions for behaviour change | Baseline and 6 months post-intervention
  Questionnaire adapted from Huijg et al. (2014) which covered the following domains: Knowledge; Skills; Social/ Professional Role & Identity; Belief about Capabilities; Optimism; Beliefs about Consequences; Intentions; GoalsAction Planning; Goals - Priorities; Memory, Attention & Decision Processes; Environmental Context & Resources; Social Influences; Emotion; Behavioural Regulation; Social & Professional Role; Work Environment. Children

CONTACTS AND LOCATIONS:
Overall Officials: Laura Basterfield, PhD, Study Director — Newcastle University
Locations (1):
- Newcastle University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This needs to be discussed with other co-authors and be checked with ethics committee from Newcastle University.

REFERENCES:
- See also: Huijg JM, Gebhardt WA, Crone MR, Dusseldorp E, Presseau J. Discriminant content validity of a theoretical domains framework questionnaire for use in implementation research. Implement Sci. 2014 Jan 15;9:11. — https://implementationscience.biomedcentral.com/articles/10.1186/1748-5908-9-11
- See also: Cole TJ, Freeman JV, Preece MA. Body mass index reference curves for the UK, 1990. Arch Dis Child. 1995 Jul;73(1):25-9 — http://www.ncbi.nlm.nih.gov/pubmed/7639544
- See also: Henderson SE, Sugden DA, Barnett AL. Movement assessment battery for children-2. Second edition (Movement ABC-2). London: The Psychological Corporation; 2007 — https://www.pearsonclinical.co.uk/Psychology/ChildCognitionNeuropsychologyandLanguage/ChildPerceptionandVisuomotorAbilities/MABC-2/MovementAssessmentBatteryforChildren-SecondEdition(MovementABC-2).aspx
- See also: Dockrell, J. (2012). Developing a communication supporting classrooms observation tool. — https://www.academia.edu/12992790/Developing_a_communication_supporting_classrooms_observation_tool